CLINICAL TRIAL: NCT04385108
Title: Identification of Predictive Immune Biomarkers Based on the Understanding of COVID-19 Pathogenesis to Influence Therapeutic Management
Brief Title: Predictive Immune Biomarkers for COVID-19 Pathogenesis
Acronym: COVIDBioToul
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/20/0162
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; COVID-19; predictive medicine; pathophysiology; immune responses
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hospitalized patients (Experimental): very well-defined population of COVID-19 patients with the following outcomes:
  * Patients with severe disease requiring on admission ICU management for ARDS,
  * Non-severe hospitalized patients with secondary clinical worsening requiring ICU management,
  * Non-severe hospitalized patients without clinical worsening requiring ICU management.
  Interventions: Biological: Blood collection on admission and longitudinally
- healthcare workers (Experimental): mildly symptomatic patients among healthcare workers attending outpatient dedicated clinics will be recruited
  Interventions: Biological: Blood collection on their first consultation and 10 to 14 days later

INTERVENTIONS:
Biological: Blood collection on admission and longitudinally — 33 mL of blood collected on admission (day 0) and longitudinally (day 4, 8 12 and in discharge)
  Arms: hospitalized patients
Biological: Blood collection on their first consultation and 10 to 14 days later — 33 mL of blood collected on their first consultation and 10 to 14 days later
  Arms: healthcare workers

SUMMARY:
The spectrum of the COVID-19 disease ranges from benign to asymptomatic to viral pneumopathy that can progress to acute respiratory distress syndrome (ARDS). The host-pathogen relationships and the physiopathological mechanisms underlying the clinical aggravation of COVID-19 patients remain misunderstood. The project aim is to create a prospective cohort of biological samples collected from well characterized COVID-19 patients. This project aims first to identify based on these samples an early immune signature predictive of clinical worsening of COVID-19 patients in order to improve their management, and secondarily to better understand pathophysiological mechanisms underlying the different phases of the disease in order to identify innovative therapeutic targets and vaccine perspectives.

DETAILED DESCRIPTION:
The World Health Organization (WHO) has recently declared pandemic the coronavirus disease 2019 (COVID-19) due to the causative severe acute respiratory syndrome (SARS) coronavirus (CoV) 2 (SARS-CoV-2). People infected with SARS-CoV-2 vary in severity from being asymptomatic to having severe pneumonia and ARDS. Predictive markers of clinical worsening after admission are lacking. Clinical deterioration often coincides with the development of host antiviral immune responses, suggesting that the inflammatory response to SARS-CoV-2 infection may underpin COVID-19 pathogenesis leading to aberrant and excessive immune responses causing lung functional disability. Relevant therapeutic strategies are still under investigation. Based on a better understanding of COVID-19 immunopathogenesis, the identification of predictive biomarkers early in the disease process would be of outstanding interest to tailor prompt therapeutic interventions.

On this basis, the project aims to create a prospective cohort of biological samples collected from COVID-19 patients followed at the Toulouse University Hospital.

This cohort will collect and cryopreserve biological samples (33 mL), including plasma and peripheral blood mononuclear cells (PBMCs), on admission (day 0) and longitudinally (day 4, 8 12 and in discharge) and will allow us to investigate our primary and secondary objectives. This cohort will be bridged with a clinical cohort in order to have a very well-defined population of COVID-19 patients with the following outcomes:

* Patients with severe disease requiring on admission intensive care unit (ICU) management for ARDS,
* Non-severe hospitalized patients with secondary clinical worsening requiring ICU management,
* Non-severe hospitalized patients without clinical worsening requiring ICU management.

In addition, mildly symptomatic patients among healthcare workers attending outpatient dedicated clinics will be recruited and blood samples will be collected on their first consultation and 10 to 14 days later in the frame of a medical surveillance program.

ELIGIBILITY:
Inclusion Criteria:

For COVID-19 hospitalized patients

* Polymerase chain reaction (PCR) proven SARS-CoV-2 infection
* Participation to Toulouse clinical cohort
* Having signed consent for inclusion in the Toulouse biobanks

For COVID-19 healthcare workers attending dedicated clinics

* PCR proven SARS-CoV-2 infection
* Having signed consent for inclusion in the Toulouse biobanks

Exclusion Criteria:

* Pregnancy or breastfeeding
* Participation in another interventional clinical study involving exploratory treatment or blood sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Immune signature | Day 0
  Analysis of the phenotypic profiling of blood T-cells by multicolor fluorescence-activated cell sorter (FACS) analysis assessing T cell subsets through the expression of a wide range of surface and intracellular markers
Dosage of cytokines and chemokines in plasma samples | Day 0
  Analysis on plasma samples of a wide range of cytokines and chemokines using multiplex

SECONDARY OUTCOMES:
Immune signature | Day 2
  Analysis of the phenotypic profiling of blood T-cells by multicolor FACS analysis assessing T cell subsets through the expression of a wide range of surface and intracellular markers
Immune signature | Day 4
  Analysis of the phenotypic profiling of blood T-cells by multicolor FACS analysis assessing T cell subsets through the expression of a wide range of surface and intracellular markers
Immune signature | Day 8
  Analysis of the phenotypic profiling of blood T-cells by multicolor FACS analysis assessing T cell subsets through the expression of a wide range of surface and intracellular markers
Immune signature | Day 12
  Analysis of the phenotypic profiling of blood T-cells by multicolor FACS analysis assessing T cell subsets through the expression of a wide range of surface and intracellular markers
Immune signature | Day 30 (or in discharge)
  Analysis of the phenotypic profiling of blood T-cells by multicolor FACS analysis assessing T cell subsets through the expression of a wide range of surface and intracellular markers
Analysis of the early dynamics of SARS-CoV-2-specific humoral immunity | Day 0
  Measurement of SARS-CoV-2 specific Immunoglobulin M, Immunoglobulin G and Immunoglobulin
Analysis of the early dynamics of SARS-CoV-2-specific humoral immunity | Day 2
  Measurement of SARS-CoV-2 specific Immunoglobulin M, Immunoglobulin G and Immunoglobulin
Analysis of the early dynamics of SARS-CoV-2-specific humoral immunity | Day 4
  Measurement of SARS-CoV-2 specific Immunoglobulin M, Immunoglobulin G and Immunoglobulin
Analysis of the early dynamics of SARS-CoV-2-specific humoral immunity | Day 8
  Measurement of SARS-CoV-2 specific Immunoglobulin M, Immunoglobulin G and Immunoglobulin
Analysis of the early dynamics of SARS-CoV-2-specific humoral immunity | Day 12
  Measurement of SARS-CoV-2 specific Immunoglobulin M, Immunoglobulin G and Immunoglobulin
Analysis of the early dynamics of SARS-CoV-2-specific humoral immunity | Day 30 (or in discharge)
  Measurement of SARS-CoV-2 specific Immunoglobulin M, Immunoglobulin G and Immunoglobulin

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MARTIN-BLONDEL, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Purpan University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dimeglio C, Herin F, Da-Silva I, Gernigon C, Porcheron M, Chapuy-Regaud S, Izopet J. Decreased Efficiency of Neutralizing Antibodies from Previously Infected or Vaccinated Individuals against the B.1.617.2 (Delta) SARS-CoV-2 Variant. Microbiol Spectr. 2022 Aug 31;10(4):e0270621. doi: 10.1128/spectrum.02706-21. Epub 2022 Jul 5. PMID 35867411
- [Derived] Dimeglio C, Herin F, Da-Silva I, Jougla I, Pradere C, Porcheron M, Martin-Blondel G, Chapuy-Regaud S, Izopet J. Heterologous ChAdOx1-S/BNT162b2 Vaccination: Neutralizing Antibody Response to Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2022 Apr 9;74(7):1315-1316. doi: 10.1093/cid/ciab705. No abstract available. PMID 34383902
- [Derived] Kreutmair S, Unger S, Nunez NG, Ingelfinger F, Alberti C, De Feo D, Krishnarajah S, Kauffmann M, Friebel E, Babaei S, Gaborit B, Lutz M, Jurado NP, Malek NP, Goepel S, Rosenberger P, Haberle HA, Ayoub I, Al-Hajj S, Nilsson J, Claassen M, Liblau R, Martin-Blondel G, Bitzer M, Roquilly A, Becher B. Distinct immunological signatures discriminate severe COVID-19 from non-SARS-CoV-2-driven critical pneumonia. Immunity. 2021 Jul 13;54(7):1578-1593.e5. doi: 10.1016/j.immuni.2021.05.002. Epub 2021 May 9. PMID 34051147